CLINICAL TRIAL: NCT05685485
Title: The Effects of Temporary Tube Ligation in Ahmed Glaucoma Valve Surgery
Brief Title: Tied Tube Trial in Glaucoma Surgery
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Glaucoma Society (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 202206072
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma Eye; Ahmed Glaucoma Valve Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Implantation: Standard Implantation
  Interventions: Procedure: Standard Implantation
- Tied off Tube: Tied off Tube
  Interventions: Procedure: Tied off Tube

INTERVENTIONS:
Procedure: Standard Implantation — Traditional Ahmed plantation without vicryl ligature
  Groups: Standard Implantation
Procedure: Tied off Tube — Ahmed implantation with vicryl ligature
  Groups: Tied off Tube

SUMMARY:
The aim of this study is to assess whether delaying early flow through the Ahmed tube shunt may improve the post-operative surgical outcomes and provide a more predictable outcome. To assess this the investigator will conduct a, randomized prospective, multi-centered study with collaborators at WashU in St. Louis, Duke University, Indiana University and the University of Pittsburgh. Participants will be randomized to have an AGV placement with tube ligation (no-early flow) and without ligation (allowing for early flow). IOP will be measured at day one, week one, and months, one, three six, and twelve. Additionally, clinical data regarding number of glaucoma medications, and complications post-operative complications will also be collected.

DETAILED DESCRIPTION:
The purpose of this study is to compare the post-operative surgical outcomes and complication rates in patients with different surgical techniques in the Ahmed FP7 glaucoma valve implant (New World Medical, Inc., Rancho Cucamonga, CA). In particular, the investigator wishes to assess whether delaying early aqueous flow by using a vicryl ligature (as done in most non-valved glaucoma drainage device implantation) will reduce the hypertensive phase, reduce early encapsulation, and optimize healing dynamics to allow for improved long term IOP results compared to standard implantation techniques.

Aggressive early aqueous flow may introduce inflammatory mediators that may increase fibrosis during wound healing. Furthermore, mechanical compression of the tissue surrounding the plate may further lead to a denser capsule and limit aqueous diffusion through Tenon's and conjunctiva. For these reasons, the investigator postulate's that the limitation of early aqueous flow through the Ahmed valve will reduce the rates of hypertensive phase, lead to a thinner and less encapsulated bleb, reduce complication rates such as hypotony, and lead to overall improvement in long-term IOP reduction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age at screening ≥ 18 years
* Inadequately controlled glaucoma or ocular hypertension
* Ahmed valve implant as the planned surgical procedure
* Patients with primary glaucomas (Primary Open Angle Glaucoma or Primary Angle Closure Glaucoma) or pseudoexfoliation, pigmentary and traumatic glaucoma with or without a previous failed trabeculectomy or other intraocular surgery.
* Primary tubes included
* Investigators to recruit consecutively all eligible patients from their clinics.
* Capable and willing to provide consent

Exclusion Criteria:

* Subjects with NLP vision
* Subjects unable/unwilling to provide informed consent
* Unavailable for regular follow up
* Previous cyclodestructive procedure
* Prior scleral buckling procedure or other external impediment to drainage device implantation
* Presence of silicone oil
* Vitreous in the anterior chamber sufficient to require a vitrectomy
* Uveitic glaucoma
* Neovascular glaucoma
* Nanophthalmos
* Patients with pathology that may cause elevated episcleral venous pressure
* Procedure combined with ocular surgery other than cataract surgery (i.e. combined tube-cataract surgery is okay)
* Any abnormality other than glaucoma in the study eye that could affect tonometry.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include patients where the clinical and surgical decision is to undergo an Ahmed glaucoma valve implantation. Participants will be identified by the ophthalmologist overseeing their glaucoma care.
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-12-18 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
IOP Change | Months 1, 3 , 6, and 12
  Change IOP

SECONDARY OUTCOMES:
Medication Change | Months 1, 3, 6, and 12
  Change glaucoma medications

OTHER OUTCOMES:
Complication Rate | Months 1, 3, 6, and 12
  Change Hypotony, Reoperations, Significant Vision Loss
Surgical Case Time | Post op day 0
  Decrease surgical case time
Capsule Thickness as measured by anterior segment OCT | month 6
  Capsule Thickness as measured by anterior segment OCT

CONTACTS AND LOCATIONS:
Overall Officials: James Liu, MD, Principal Investigator — Washington University St. Louis MO
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No